CLINICAL TRIAL: NCT03780465
Title: A Single Centre Study of Pharmacokinetics and Safety of NOX66 in Healthy Subjects
Brief Title: A Study of Safety and Tolerability of NOX66 in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to obtain PK data at a later date
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NOX66-003
Record Dates: First submitted 2018-12-05; First posted 2018-12-19 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The pharmacist preparing the study medication and the study nurse administering the study medication are not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral idronoxil (Active Comparator): 10 male and female subjects randomised to 400 mg active Oral idronoxil suspension or oral placebo suspension (n=8 active; n= 2 placebo).
  Interventions: Drug: Oral idronoxil suspension
- NOX66 400 mg (Experimental): 10 male and female subjects randomised to 400 mg active NOX66 (A) suppository or 400 mg active NOX66 (B) suppository or suppository placebo (n=8 active; n= 2 placebo).
  Interventions: Drug: NOX66 (A); Drug: NOX66 (B)
- NOX66 600 mg (Experimental): 10 male and female subjects randomised to 600 mg active NOX66 (A) suppository or 600 mg active NOX66 (B) suppository or suppository placebo (n=8 active; n= 2 placebo).
  Interventions: Drug: NOX66 (A); Drug: NOX66 (B)

INTERVENTIONS:
Drug: Oral idronoxil suspension — Idronoxil powder up to 150 ml ORA-BLEND® flavoured syrup
  Arms: Oral idronoxil
Drug: NOX66 (A) — Idronoxil formulated in suppository base A
  Arms: NOX66 400 mg; NOX66 600 mg
Drug: NOX66 (B) — Idronoxil formulated in suppository base B
  Arms: NOX66 400 mg; NOX66 600 mg

SUMMARY:
A Phase 1, double- blinded, randomised, placebo-controlled study to assess safety, tolerability and pharmacokinetics of 2 formulations of NOX66 in healthy subjects when administered over 4 cohorts as single NOX66 dose of 400 mg and 600 mg in comparison to single oral dose of 400 mg idronoxil.

DETAILED DESCRIPTION:
The study will be a single-centre study of NOX66 in two formulations administered once rectally and oral idronoxil . Approximately 50 subjects will be enrolled in 5 cohorts, comprising 1 oral dose (400 mg) and 4 NOX66 dose Cohorts (400 and 600 mg in formulation A and B).

Eligible subjects will be admitted to the research clinic the day prior to dosing for baseline evaluations and will be fasted for a minimum of 10 hours prior to pre-dosing procedures. On treatment day, subjects will be administered NOX66 suppository as single dose or as oral suspension. Subjects remain in the clinic for 24 hours (h) after each dose for safety and pharmacokinetic assessments and return for 3 follow up visits.

Ten subjects will be assigned to treatment dose Cohorts (1-5) and subjects within each of these cohorts will be randomised to either active or placebo (n=8 active; n= 2 placebo).

For all dose cohorts, there will be two sentinel subjects (2 active) who will be dosed at a minimum 24 hours prior to remainder of the cohort who will be dosed simultaneously thereafter. Dose escalation of NOX66 dose cohorts to occur once safety and PK has been confirmed, by Data Safety Monitoring Board, in subjects in the prior cohort as applicable.

Following interim review of accumulating PK data from first 3 cohorts, the Sponsor may modify subject numbers within a cohort or cohort dose levels and implemented following approval by IRB.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Male and/or female subjects, 18 - 55 years of age.
3. BMI of 17.5 to 30 kg/m2 and a total body weight >50 kg.
4. Negative hepatitis panel (including HBsAg and anti-HCV) and negative HIV antibody screens.
5. Negative test for selected drugs of abuse.
6. Males and females of childbearing potential who are not abstinent from heterosexual intercourse as part of their usual and preferred lifestyle must agree for the study duration and for 3 months after study to use two effective means of contraception (hormonal contraception, intrauterine device, condoms). Surgical sterilisation >3 months prior to Screening is acceptable.

   * Postmenopausal females should have menopause confirmed by follicle-stimulating hormone (FSH) testing.
   * Subjects who have same sex partners or who practice abstinence in line with standard and preferred lifestyle will not be required to use contraception.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated asymptomatic, penicillin, seasonal allergies at the time of dosing).
2. 12-lead ECG at screening or at first admission to the study center. Subjects with a QTcF interval >450 msec or QRS interval ≥110 msec will be excluded.
3. Treatment with an investigational drug /device within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer).
4. Other severe acute or chronic medical or psychiatric conditions or a laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the principal investigator (PI), would make the subject inappropriate for entry into this study.
5. Abnormal nutritional status, including unconventional and abnormal dietary habits; excessive or unusual vitamin intake; malabsorption (oral cohort only).
6. Has history of significant drug or alcohol abuse within past 5 years or has a positive drug screen.
7. Smoking or use of nicotine-containing substances within past 2 months with the exception for social smokers who will be allowed a maximum of 5 cigarettes per week.
8. Has use of any prescription or nonprescription medications or herbal supplements, except for paracetamol, within 14 days before the first dose of study drug, unless approved by the PI and sponsor.
9. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy, cholecystectomy, and hernia repair will be allowed.
10. Consumption of grapefruit/starfruit-containing foods and beverages or other CYP3A4 inhibitors or inducers for 72 hours prior to Screening and during the entire study.
11. Donation of blood from 30 days prior to Screening through Study Completion/End of treatment (ET), inclusive, or plasma from 2 weeks prior to Screening through Study Completion/ET, inclusive.
12. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.
13. Use of alcohol within previous 24 hours or use of caffeine within previous 12 hours of Day -1 admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Area Under the concentration-time Curve for idronoxil from NOX66 and oral formulations | Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
  AUC will be determined form blood plasma and urine taken at pre-dose and post dose time points..
  Plasma concentration data for idronoxil will be summarised for the PK population by treatment and scheduled sampling time.
Maximal observed concentration for idronoxil levels from NOX66 and oral formulations | Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
  Maximal observed concentration of idronoxil will be assessed from blood plasma taken at pre-dose and post dose time points .
Time to reach maximum observed concentration from idronoxil for NOX66 formulations and oral | Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
  Time to occurrence of maximum observed concentration will be measured from blood plasma taken at pre-dose and post dose time points.
Terminal half-life of Plasma and Urine idronoxil from NOX66 and oral formulations and oral | Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose.
  Apparent terminal half-life will be assessed from blood plasma and urine taken at pre-dose and post dose time points.
Total body clearance of idronoxil after administration of NOX66 and oral formulations | Day 1 pre-dose and at multiple time points (up to 144 hours) post-dose
  Total body clearance will be assessed from blood plasma and urine taken at pre-dose and post dose time points.

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events | From screening up to end of study (144 hours)
  Safety and tolerability of single doses of NOX66 formulations by assessing adverse events according to CTCAE version 5.0
Relative bioavailability of NOX66 formulations compared to the oral idronoxil | From pre-dose up to end of study (144 hours)
  To compare area under the concentration curve (AUC) of idronoxil from NOX66 to orally administered idronoxil.
Number subjects with clinical significant ECGs | Telemetry 10 hours prior dosing continuously for 24 hours post dosing (cohorts 1, 4 and 5); safety ECGs for all cohorts pre dose and post dose to 144 hrs or end of study.
  Continuous cardiac monitoring by telemetry Holter device for oral dose cohort 1 and highest NOX66 dose cohorts (4 and 5) and safety ECGs for all dose cohorts.
Number subjects with clinical significant abnormalities in lab tests | Screening to 7 days
  Routine safety labs for all cohorts
Number subjects with clinical significant abnormalities in vital signs | Screening to 7 days
  Routine vital signs for all cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Marinella Messina, PhD, Study Chair — Noxopharm Limited
Locations (1):
- Nucleus Network Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measure will be made available within 12 months after study completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after study completion